CLINICAL TRIAL: NCT02111759
Title: The Effect of Knee Flexion Angle for Graft Fixation During Single-Bundle Anterior Cruciate Ligament Reconstruction - A Multicentre, Patient and Assessor Blinded, Stratified, Two-arm Parallel Group Superiority Trial
Brief Title: The Effect of Knee Flexion Angle for Graft Fixation During Single-Bundle Anterior Cruciate Ligament Reconstruction
Acronym: FIRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto Orthopaedic Sports Medicine (Other)
Collaborators: Arthroscopy Association of North America (Other)
Responsible Party: Principal Investigator, Jaskarndip Chahal, Principal Investigator, University of Toronto Orthopaedic Sports Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTOSM0001
Record Dates: First submitted 2014-03-27; First posted 2014-04-11 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- knee flexion angle 2 (Other): 30 degrees of knee flexion during ACL graft fixation
  Interventions: Procedure: knee flexion angle 2
- knee flexion angle 1 (Other): 0 degrees of knee flexion during ACL graft fixation
  Interventions: Procedure: knee flexion angle 1

INTERVENTIONS:
Procedure: knee flexion angle 1 — 0 degrees of knee flexion during ACL graft fixation
  Arms: knee flexion angle 1
Procedure: knee flexion angle 2 — 30 degrees of knee flexion during ACL graft fixation
  Arms: knee flexion angle 2

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to determine if the knee flexion angle (KFA) during anterior cruciate ligament reconstruction (ACLR) graft fixation has an effect on postoperative outcomes. The specific research questions are: what is the effect of the KFA on 1) patient-reported outcomes; 2) postoperative extension loss; 3) antero-posterior (AP) knee stability; 4) rate of re-operation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients older than 16 years old with an isolated anterior cruciate ligament injury as diagnosed by clinical examination and MRI
* No pre-existing arthritis as defined by the Kellgren-Lawrence radiographic rating system
* Patients treated with an initial period of rehabilitation to eliminate swelling, optimize quadriceps strength and restore range of motion
* surgical management with a transtibial or anteromedial portal single-bundle ACLR with bone patella tendon bone (BPTB) autograft by a fellowship-trained sports medicine surgeon.

Exclusion Criteria:

* Acute ACL injuries that have not undergone an initial period of physical therapy in order to restore the aforementioned parameters
* Associated grade III injury to the MCL (medial opening >10mm at 30 degrees of knee flexion or any medial opening in extension)
* Presence of a PCL or posterolateral corner injury
* Lack of informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 24 months postoperatively

SECONDARY OUTCOMES:
KOOS scores | 3, 6, and 12 months
Marx Activity Score (MAS) | 3, 6, 12, 24 months
the degree of extension loss in the affected knee (vs. contralateral knee) | 3, 6, 12, and 24 months
  the degree of extension in the affected knee as measured by a goniometer
Side to side differences in anterior-posterior (AP) stability | 3, 6, 12, and 24 months
  differences in anterior-posterior knee (in the affected knee vs. the contralateral knee) as measured by the KT1000 arthrometer

CONTACTS AND LOCATIONS:
Overall Officials: Jaskarndip Chahal, MD, Principal Investigator — University of Toronto Orthopaedic Sports Medicine
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada